CLINICAL TRIAL: NCT06618911
Title: Evaluation of the Efficacy of Electroacupuncture in the Treatment of Functional Dyspepsia: A Pilot Study
Brief Title: Evaluation of the Efficacy of Electroacupuncture in the Treatment of Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Liang (Other)
Collaborators: Zhejiang Provincial Department of Science and Technology (Unknown)
Responsible Party: Sponsor-Investigator, Yi Liang, Research Fellow, The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240903074110247
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Functional Dyspepsia
Keywords: electroacupuncture; functional dyspepsia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5 Hz Electroacupuncture Group (Experimental): Participants will receive electroacupuncture at a frequency of 5 Hz at four acupoints: Liangmen (ST21) and Tianshu (ST25) (local acupoints), and Zusanli (ST36) and Xiajuxu (ST39) (distal acupoints). Disposable needles will be inserted until the "deqi" sensation is achieved. The needles will be connected to an SDZ-IIB electroacupuncture device set at 5 Hz, with stimulation lasting 30 minutes per session. Participants will receive 3 sessions per week for 4 weeks (total: 12 sessions). This group aims to evaluate the efficacy of low-frequency electroacupuncture for treating functional dyspepsia.
  Interventions: Other: 5 Hz electroacupuncture
- 100 Hz Electroacupuncture Group (Experimental): Participants will receive electroacupuncture at a frequency of 100 Hz at the same four acupoints: Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39). Needles will be inserted to induce the "deqi" sensation and connected to an SDZ-IIB device set at 100 Hz, with stimulation lasting 30 minutes per session. Participants will receive 3 sessions per week for 4 weeks (total: 12 sessions). This group assesses the efficacy of high-frequency electroacupuncture for functional dyspepsia.
  Interventions: Other: 100 Hz electroacupuncture
- Sham Electroacupuncture (Control) Group (Sham Comparator): Participants will receive sham electroacupuncture at the same acupoints: Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39). Non-penetrating needles will touch the skin but will not induce "deqi." A sham electroacupuncture device (no actual current) will be used, and treatment will last 30 minutes per session. Participants will receive 3 sessions per week for 4 weeks (total: 12 sessions). This arm serves as a placebo control to evaluate the true effect of electroacupuncture.
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: 5 Hz electroacupuncture — Intervention Description:
  The intervention in this study involves the use of electroacupuncture (EA), a combination of traditional acupuncture and electrical stimulation.
  Acupoints Selection: Electroacupuncture will be performed at specific acupoints associated with the stomach and digestive system. The local acupoints chosen are Liangmen (ST21) and Tianshu (ST25), while the distal acupoints are Zusanli (ST36) and Xiajuxu (ST39). This selection is based on Traditional Chinese Medicine (TCM) principles for treating functional dyspepsia.
  Frequency: 5 Hz
  Arms: 5 Hz Electroacupuncture Group
Other: Sham electroacupuncture — Participants will receive sham electroacupuncture at the same acupoints: Liangmen (ST21), Tianshu (ST25), Zusanli (ST36), and Xiajuxu (ST39). Non-penetrating needles will touch the skin but will not induce "deqi." A sham electroacupuncture device (no actual current) will be used, and treatment will last 30 minutes per session. Participants will receive 3 sessions per week for 4 weeks (total: 12 sessions). This arm serves as a placebo control to evaluate the true effect of electroacupuncture.
  Arms: Sham Electroacupuncture (Control) Group
Other: 100 Hz electroacupuncture — Intervention Description:
  The intervention in this study involves the use of electroacupuncture (EA), a combination of traditional acupuncture and electrical stimulation.
  Acupoints Selection: Electroacupuncture will be performed at specific acupoints associated with the stomach and digestive system. The local acupoints chosen are Liangmen (ST21) and Tianshu (ST25), while the distal acupoints are Zusanli (ST36) and Xiajuxu (ST39). This selection is based on Traditional Chinese Medicine (TCM) principles for treating functional dyspepsia.
  Frequency: 100 Hz
  Arms: 100 Hz Electroacupuncture Group

SUMMARY:
Brief Summary Template for the Study:

The goal of this clinical trial is to evaluate whether electroacupuncture can treat functional dyspepsia (FD) in adult participants aged 18 to 65 years, including both males and females, who have been diagnosed with functional dyspepsia based on the Rome IV criteria. The main questions it aims to answer are:

* Does 5 Hz electroacupuncture improve symptoms in functional dyspepsia patients?
* Does 100 Hz electroacupuncture improve symptoms in functional dyspepsia patients?
* Are there differences in the efficacy between 5 Hz and 100 Hz electroacupuncture in treating functional dyspepsia and its subtypes (PDS and EPS)?

Researchers will compare the effects of 5 Hz electroacupuncture, 100 Hz electroacupuncture, and sham electroacupuncture to determine which approach provides more significant symptom relief and whether different frequencies have varying impacts on FD subtypes.

Participants will:

* Receive electroacupuncture treatment at specific acupoints (such as Liangmen, Tianshu, Zusanli, and Xiajuxu) for 30-minute sessions, 3 times a week for 4 weeks.
* Be randomly assigned to one of the following groups: 5 Hz electroacupuncture, 100 Hz electroacupuncture, or sham electroacupuncture (control).
* Have their functional dyspepsia symptoms, quality of life, and any adverse effects monitored and evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with functional dyspepsia based on Rome IV diagnostic criteria.
* Aged 18 to 80 years, inclusive, with no gender restrictions.
* Normal endoscopy results within the past year, showing no structural explanation for symptoms.
* No acupuncture treatment in the last month.
* Not participating in any other clinical trials in the past 2 months.
* Able to understand and provide informed consent.

Exclusion Criteria:

* Presence of serious or malignant diseases (e.g., cirrhosis, heart failure, gastrointestinal tumors) that could explain dyspepsia symptoms.
* Positive for Helicobacter pylori infection based on C-13 urea breath test or gastric biopsy.
* History of gastrointestinal surgery (excluding laparoscopic and other minimally invasive surgeries).
* Recent use (within 2 weeks) of medications affecting dyspepsia, including prokinetics, proton pump inhibitors, antacids, or antidepressants.
* Presence of severe mental or physical conditions, such as dementia or illiteracy, that could interfere with study participation.
* Severe coagulation disorders.
* Substance abuse or alcohol dependence.
* Pregnant or breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-04-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Symptom Improvement Rate at Week 4 | 4 weeks after the start of treatment.
  The primary outcome is the percentage of participants experiencing symptom improvement using the 7-point Likert scale for Overall Treatment Effect (OTE).
  The Overall Treatment Effect (OTE) questionnaire was categorized as "extremely worse than baseline," "worse than baseline," "slightly worse than baseline," "no change," "slightly improved than baseline," "improved than baseline," or "much improved than baseline."
  Participants will rate their symptom severity compared to baseline, and those reporting "improved than baseline" or "much improved than baseline"will be considered responders.
  The primary outcome will assess the efficacy of 5 Hz and 100 Hz electroacupuncture compared to sham treatment.
Main Symptom Resolution Rate at Week 4 | 4 weeks after the start of treatment.
  The second primary outcome is the rate of complete resolution of the main symptoms of functional dyspepsia at week 4. For Postprandial Distress Syndrome (PDS), the primary symptoms are postprandial fullness and early satiety; for Epigastric Pain Syndrome (EPS), the main symptoms are epigastric pain and burning. Complete resolution is defined as a score of 0 for the respective main symptoms on a validated symptom severity scale.
  The severity of each symptom is divided into: no symptoms (0 points), mild (1 point), moderate (2 points), and severe (3 points).
  The outcome will compare the resolution rates between the 5 Hz, 100 Hz, and sham electroacupuncture groups.

SECONDARY OUTCOMES:
Global Overall Symptom (GOS) Score Change | Baseline to Week 4
  The Global Overall Symptom (GOS) score assesses eight symptoms associated with functional dyspepsia (e.g., epigastric pain, burning, fullness, early satiety, nausea, bloating). Scores range from 1 (no problem) to 7 (very severe problem).
  Scoring is as follows: 1 = no problem (no symptoms); 2 = minimal problem (can be easily ignored); 3 = mild problem (can be ignored with effort); 4 = moderate problem (cannot be ignored, but does not interfere with daily activities); 5 = moderately severe problem (cannot be ignored, occasionally limits daily activities); 6 = severe problem (cannot be ignored, often limits concentration on daily activities); 7 = very severe problem (cannot be ignored, severely limits daily activities.
  The change from baseline to week 4 will be compared between the 5 Hz, 100 Hz, and sham electroacupuncture groups.
Nepean Dyspepsia Index (NDI) Score Change | Baseline to Week 4
  The Nepean Dyspepsia Index (NDI) evaluates the impact of dyspepsia on patients &amp;amp;#39;quality of life across five domains (e.g., tension, interference with daily activities). The change in NDI score from baseline to week 4 will be used to assess the efficacy of the interventions in improving quality of life.
  Higher scores on the Nepean Dyspepsia Index (NDI) indicate more severe symptoms
Hospital Anxiety and Depression Scale (HADS) Score Change | Baseline to Week 4
  The Hospital Anxiety and Depression Scale (HADS) measures levels of anxiety and depression, which are often associated with functional dyspepsia. Changes in HADS scores from baseline to week 4 will be evaluated to determine if electroacupuncture has an impact on emotional well-being.
  The scores of anxiety and depression subscales are divided into: 0-7 points for no symptoms; 8-10 points for suspected presence; 11-21 points for definite presence; When scoring, 8 points is the starting point, that is, both suspected and symptomatic are positive.
Treatment Expectation Score | Prior to the first treatment (Baseline)
  Participants&amp;amp;amp;amp;amp;amp;#39; expectations regarding the effectiveness of electroacupuncture will be assessed using a 5-point Likert scale (e.g., strongly agree to strongly disagree) prior to the first treatment. This outcome will be used to determine the role of treatment expectations in the perceived efficacy of electroacupuncture.
Blind evaluation | immediately after 1st and 6th treatment sessions
  Participants perception of whether they received real or sham electroacupuncture will be assessed after the 1st and 6th treatment sessions to evaluate the effectiveness of blinding in the sham group.

OTHER OUTCOMES:
Subgroup Analysis of Symptom Improvement by FD Subtypes (PDS vs. EPS) | At Week 4
  This outcome will assess whether the efficacy of 5 Hz and 100 Hz electroacupuncture differs between patients with Postprandial Distress Syndrome (PDS) and Epigastric Pain Syndrome (EPS). The primary and secondary outcome measures (symptom improvement, main symptom resolution, and quality of life scores) will be analyzed separately for these two subgroups. The comparison aims to determine if electroacupuncture has varying levels of effectiveness depending on the functional dyspepsia subtype.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The Third Affiliated Hospital of Zhejiang Chinese Medicinal University, Hangzhou, None Selected
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF